CLINICAL TRIAL: NCT00005990
Title: Phase I and Pharmacokinetic Study of the Farnesyl Transferase Inhibitor, R115777, in Combination With Topotecan
Brief Title: R115777 Plus Topotecan in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000067979; NYU-9932; NCI-T99-0110
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2006-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — tipifarnib; Topotecan

INTERVENTIONS:
Drug: tipifarnib
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of R115777 plus topotecan in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the dose-limiting toxic effects of R115777 and topotecan in patients with advanced solid tumors.
* Determine the maximum tolerated dose of this regimen in these patients.
* Determine pharmacokinetic profiles of topotecan alone and in combination with R115777 in these patients.
* Measure the inhibition of ras-farnesylation and topo-1 inhibition in peripheral blood mononuclear cells in these patients when treated with this regimen.
* Determine activity of this treatment in these patients.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive oral R115777 twice daily on days 2-21 (in the first course only R115777 begins on day 3) and topotecan IV continuously on days 1-21. Treatment continues every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of R115777 and topotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 3 or 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 18-24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced solid tumor not amenable to standard curative therapy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* At least 6 months

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* SGOT no greater than 5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 5 times ULN
* No significant hepatic dysfunction that would preclude study

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 50 mL/min

Cardiovascular:

* No significant cardiovascular dysfunction that would preclude study

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No malabsorption syndrome, partial or complete bowel obstruction, disease significantly affecting gastrointestinal function, or major resection of the stomach or proximal small bowel
* At least 1 week since prior active infection requiring systemic medical therapy
* No significant organ system dysfunction (neurologic, endocrine) that would preclude study
* No dementia or altered mental status that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No more than 3 prior chemotherapy regimens
* At least 4 weeks since prior chemotherapy and recovered

Endocrine therapy:

* Not specified

Radiotherapy:

* No more than 25% of bone marrow volume irradiated
* No prior pelvic radiation
* At least 4 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Primary Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard S. Hochster, MD, Study Chair — NYU Langone Health
Locations (1):
- NYU Cancer Institute at New York University Medical Center, New York, New York, United States